CLINICAL TRIAL: NCT06599476
Title: Use of Rectal Spacers in Prostate Cancer Patients Undergoing Radiation Therapy: a Prospective Clinical Study
Brief Title: Rectal Spacers in Prostate Cancer Patients Undergoing Radiation Therapy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Advanced Radiation Centers of New York (Other)
Responsible Party: Principal Investigator, Shawn Zimberg, MD, Dr Shawn Zimberg, Radiation Oncology Medical Director, Radiation Oncology, Advanced Radiation Centers of New York
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 1372621
Record Dates: First submitted 2024-08-26; First posted 2024-09-19 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2024-08

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- BioProtect Balloon Implant System (Experimental): The Bio Protect Balloon Implant System (BioProtectLtd.,TzurYigal,Israel) is an Food and Drug Administration approved rectal spacer that consists of a solid biodegradable balloon-shaped material composed of poly L-Lactide-co-caprolactone
  Interventions: Device: BioProtect Balloon Implant™ System

INTERVENTIONS:
Device: BioProtect Balloon Implant™ System — The BioProtect Balloon Implant System is intended to temporarily position the anterior rectal wall away from the prostate during radiotherapy for prostate cancer, and by creating this space, to reduce the radiation dose delivered to the anterior rectum. The balloon is inserted into the perirectal space and inflated to its pre-defined size. The Balloon is made of biodegradable materials that maintain the space for the entire course of prostate radiation treatment and are absorbed by the patient's body over time

SUMMARY:
This is a prospective clinical study involving up to 150 subjects with localized prostate cancer who are scheduled for radiation treatment with rectal spacer placement.

The goal of this clinical trial is to assess the safety and efficacy of perirectal spacers in patients undergoing radiation therapy for the treatment of localized prostate cancer.

Study visits:

* Screening
* Spacer placement
* Treatment planning simulation
* End of the radiation treatment
* 1,3,and 6-months FU visits.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with prostate cancer ≥ 18 years of age.
2. Patients are in one of the following risk groups:

   * T1-T3 prostate cancer with no posterior extra capsular extension
   * Gleason score ≤ 7
3. Planned for radiation treatment with rectal spacer.
4. Ability to understand and the willingness to sign a written informed consent form.

Exclusion Criteria:

1. Metastatic disease.
2. Previously treated localized adenocarcinoma of the prostate.
3. Active Inflammatory bowel disease requiring treatment with steroids.
4. Prior total prostatectomy.
5. Current urinary tract infection.
6. Acute or chronic prostatitis.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-05-21 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Dosimetry | 6 months
  Dose-volume histogram (DVH) including the percent of the rectal volume receiving 70 Gy

CONTACTS AND LOCATIONS:
Locations (1):
- Advanced Radiation Centers of New York, New Hyde Park, New York, United States